CLINICAL TRIAL: NCT04939441
Title: Regression of Liver Fibrosis by Tenofovir Alafenamide (TAF) in Treatment-Naive CHB Related Fibrosis/Cirrhosis: a 96w Open-label Multicenter Study
Brief Title: Regression of Liver Fibrosis by Tenofovir Alafenamide (TAF)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jidong Jia (Other)
Collaborators: Beijing Ditan Hospital (Other); ShuGuang Hospital (Other); Tianjin Third Central Hospital (Other); Huashan Hospital (Other); The Sixth Peoples Hospital of Zhengzhou (Unknown); Tianjin Second People's Hospital (Other); Ruijin Hospital (Other); Shanghai East Hospital (Other)
Responsible Party: Sponsor-Investigator, Jidong Jia, Director of Liver Research Center, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-CN-320-5613
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; Liver fibrosis, Liver cirrhosis; Tenofovir alafenamide
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Cirrhosis | interventions — tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Subjects will be treated for 96 weeks with TAF [Vemlidy® 25mg QD] monotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAF group (Experimental): TAF [Vemlidy® 25mg QD] monotherapy
  Interventions: Drug: Tenofovir alafenamide

INTERVENTIONS:
Drug: Tenofovir alafenamide — Subjects will be treated for 96 weeks with TAF [Vemlidy® 25mg QD] monotherapy
  Other Names: Vemlidy®

SUMMARY:
Tenofovir alafenamide (TAF) is a new prodrug of tenofovir developed to treat patients with chronic hepatitis B virus (HBV) infection. Whereas, the long-term effect of TAF to liver fibrosis is still unknown. Here, we enrolled treatment naive CHB patients with biopsy-proven significant fibrosis (METAVIR fibrosis stage ≥ F2). All enrolled subjects will be treated with TAF monotherapy for 96 weeks. After 96 weeks of therapy, the second liver biopsy will be performed to evaluate the rate of liver fibrosis regression. During this study, all subjects will be assessed for laboratory tests, imaging examination at baseline, first 12-week and every 24-week during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18-69 years old (inclusive);
* BMI (18-30 kg/m2);
* Chronic hepatitis B virus (HBV) infection, defined as positive serum hepatitis B s-antigen (HBsAg) for more than 6 months; or chronic hepatitis B proven by live biopsy;
* Not received nucleoside (acid) analogue and/or interferon therapy (treatment-naive);
* Liver biopsy performed within 6 months before treatment and had readable biopsy slides or agrees to have a biopsy performed prior to baseline;
* METAVIR fibrosis stage ≥ F2;
* For patients without cirrhosis (F2/3), HBV DNA levels >2000 IU/mL before treatment; For patients with cirrhosis (F4), HBV DNA >20 IU/mL before treatment;
* ALT≤10 ULN before treatment;
* Creatinine clearance ≥ 50 mL/min;
* Agreement not to undertake other HBV systemic antiviral or interferon (IFN) regimens during participation in this study;
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Patients with Child-Turcotte-Pugh（CTP）score ≥ 7;
* Patients with decompensated cirrhosis: including ascites, hepatic encephalopathy, esophageal varices bleeding or other complications of decompensated cirrhosis or liver transplantation;
* Patients co-infection with hepatitis C virus (HCV), human immunodeficiency virus (HIV), or hepatitis delta virus (HDV), or alcoholic liver diseases, autoimmune liver disease, genetic liver disease, drug-induced liver injury, non-alcoholic fatty liver disease or other chronic liver diseases;
* Patients with evidence of hepatocellular carcinoma (HCC) by imaging with or without AFP;
* Patients with other uncured malignant tumors;
* Patients with organ or bone marrow transplantation;
* Patients currently receiving therapy with immunomodulators (eg, corticosteroids, etc.), investigational agents, nephrotoxic agents, or agents susceptible of modifying renal excretion;
* Patients who are allergic to any component of TAF;
* Patients who recently or newly started bisphosphate (within 1 month);
* Patients with active alcohol or drug abuse or history of alcohol or drug abuse (hinder compliance with treatment, or participation in the study or interpretation of results considered by the Investigator);
* Patients with significant renal, cardiovascular, pulmonary, or neurological disease
* Males and females of reproductive potential who are unwilling to use an effective method of contraception during the study;
* Pregnant women, women who are breast feeding or who believe they may wish to become pregnant during the course of the study;
* Not suitable for this study identified by researchers.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with fibrosis regression | Week 96
  Fibrosis stage decrease at least 1 point by Ishak score or "Predominantly Regressive" by "Beijing classification"
HBV DNA undetectable rate | Week 96
  Serum HBV DNA <20 IU/mL

SECONDARY OUTCOMES:
Percentage of liver stiffness decrease >= 30% | Week 48 and Week 96
  Proportion of patients with liver stiffness decrease >= 30% from baseline to week 48 and 96
HBV DNA undetectable rate | Week 24, Week 48 and Week 72
  HBV DNA undetectable rate at week 24, 48, and 72
ALT normalization rate | Week 48 and Week 96
  Proportion of patients with ALT <= 1.0xULN
HBeAg and HBsAg loss and seroconversion rate | Week 48 and Week 96
  Proportions of patients with HBsAg loss and seroconversion to anti-HBs, and proportions of patients with HBeAg loss and seroconversion to anti-HBe.
Changes in renal function | Week 48 and Week 96
  Changes of eGFR (estimated Glomerular Filtration rate) from baseline to week 48 and 96
Changes of bone mineral density | Week 48 and Week 96
  Percentage changes in spine BMD and hip BMD from baseline to week 48 and 96
Incidence of liver-related endpoint events | Week 96
  liver-related endpoint events: decompensation, HCC, liver transplantation, liver-related death

CONTACTS AND LOCATIONS:
Overall Officials: Jidong Jia, Principal Investigator — Beijing Friendship Hospital, Capital Medical Hospital
Locations (7):
- China (7):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Shuguang Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Result] Chan HL, Fung S, Seto WK, Chuang WL, Chen CY, Kim HJ, Hui AJ, Janssen HL, Chowdhury A, Tsang TY, Mehta R, Gane E, Flaherty JF, Massetto B, Gaggar A, Kitrinos KM, Lin L, Subramanian GM, McHutchison JG, Lim YS, Acharya SK, Agarwal K; GS-US-320-0110 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of HBeAg-positive chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):185-195. doi: 10.1016/S2468-1253(16)30024-3. Epub 2016 Sep 22. PMID 28404091
- [Result] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092
- [Result] Agarwal K, Brunetto M, Seto WK, Lim YS, Fung S, Marcellin P, Ahn SH, Izumi N, Chuang WL, Bae H, Sharma M, Janssen HLA, Pan CQ, Celen MK, Furusyo N, Shalimar D, Yoon KT, Trinh H, Flaherty JF, Gaggar A, Lau AH, Cathcart AL, Lin L, Bhardwaj N, Suri V, Mani Subramanian G, Gane EJ, Buti M, Chan HLY; GS-US-320-0110; GS-US-320-0108 Investigators. 96 weeks treatment of tenofovir alafenamide vs. tenofovir disoproxil fumarate for hepatitis B virus infection. J Hepatol. 2018 Apr;68(4):672-681. doi: 10.1016/j.jhep.2017.11.039. Epub 2018 Jan 17. PMID 29756595